CLINICAL TRIAL: NCT06214663
Title: Investigation of the Analgesic Effects of Intradermal and Subdermal Sterile Water Injection on Active Labor Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: E2-20-11
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Labor Pain and to Reduce Pain
Keywords: Delivery; Pain; Analgesia
MeSH Terms: conditions — Labor Pain; Pain; Agnosia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients in active labor (6 cm cervical dilatation) will be randomly divided into 3 groups. For each patient, first, VAS score (visual analogue scale: patients were asked to evaluate their own pain on a vertical, unnumbered scale. Then, the patient's evaluation was graded with the help of a scale divided into 1/10 sections of the same length as the scale: "0: no pain and 10: "unbearable pain") will be measured for labor pain and repeated at 10, 30, 60 and 90 minutes after injection. Injections will be administered over the sacral area (both posterior iliac spines and 2 cm downward and medial), and this technique was described by Lytzen et al in 1989 and later standardized. The results will be compared between the three groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 0.9 NaCl solution — Saline injections will be administered over the sacral area (both posterior iliac spines and 2 cm downward and medial), and this technique was described by Lytzen et al in 1989 and later standardized. The results will be compared between the three groups.

SUMMARY:
Labour pain has different locations, intensity, quality and meaning for each woman, and the experience of pain changes throughout the delivery process. This pain is often associated with varying degrees of fetal malposition, particularly occipito-posterior position, which may apply pressure on pain-sensitive structures within the pelvis. Administration of Injections into the sacral area (both posterior iliac spines and 2 cm downward and medial) is used and have been shown to relieve the pain of labor. Controlling pain with simple methods can reduce the desire of mothers to give birth by cesarean section and make them more diligent for normal birth.

The benefit we expect from the research; Since sterile water injection is a safe, effective and low-cost method, it is important to understand the effectiveness of its use to reduce labor pain. It also aims to increase the knowledge of gynecologists about this method.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women with cephalic presentation who are admitted to the delivery room clinic for delivery, who do not have an additional chronic disease, who have not given birth before, and who are in the second stage of labor (active cervical dilatation of 6 cm and above) will be included in the study.

Exclusion Criteria:

* Patients who do not volunteer to participate in the study will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women
Enrollment: 30 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Investigation of the analgesic effects of intradermal and subdermal sterile water injection on active labor pain. | 10, 30, 60 and 90 minutes after injection
  The benefit we expect from the research; Since sterile water injection is a safe, effective and low-cost method, it is important to understand the effectiveness of its use to reduce labor pain.
  he patient's (in active labor with 6 cm cervical dilatation) VAS score evaluation will be measured for labor pain and repeated.

IPD SHARING:
Plan to Share IPD: Undecided